CLINICAL TRIAL: NCT04524975
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding, Pilot Study to Assess the Efficacy and Safety of CD-008-0045 in Patients With Generalized Anxiety Disorder
Brief Title: А Dose-finding Study to Assess the Efficacy and Safety of CD-008-0045 in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ChemRar Research and Development Institute, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS-CD0080045-04
Record Dates: First submitted 2020-08-15; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorder Generalized
Keywords: Anti-Anxiety Agents; Anxiety Disorder Generalized
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled, dose-ranging pilot study to assess the efficacy and safety of CD-008-0045 in patients with GAD. The primary study objective is to select the dosage regimen for CD-008-0045 (20 mg BID or TID) based on preliminary assessment of its efficacy versus placebo according to frequency of treatment response at Week 8 in patients with GAD. Treatment response is considered as ≥ 50% decrease of the Hamilton Anxiety Rating Scale (HARS) total score from baseline.
Who Masked: Participant, Investigator
Masking Description: Dose blinding will be performed using Placebo. Patient will receive 3 vials labeled for study drug administration as follows: 1 capsule in the morning, afternoon, and evening.
  Package numbers were assigned via IWRS. Thus, during the Study Treatment period, neither the patient nor the Investigator knew the group to which the patient was allocated. Single blinding was performed during the Placebo Run-in and Follow-up periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CD-008-0045 60 mg/day (Experimental): Patients assigned to the CD-008-0045 60 mg/day group will receive 1 capsule of CD-008-0045 (20 mg) before breakfast, lunch, and dinner for 8 weeks
  Interventions: Drug: CD-008-0045
- CD-008-0045 40 mg/day (Experimental): Patients assigned to the CD-008-0045 40 mg/day group will receive 1 capsule of CD-008-0045 (20 mg) before breakfast and before dinner, and 1 placebo capsule before lunch for 8 weeks.
  Interventions: Drug: CD-008-0045; Drug: Placebo
- Placebo (Placebo Comparator): Patients assigned to the Placebo group will receive 1 placebo capsule before breakfast, lunch, and dinner for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD-008-0045 — CD-008-0045 20 mg capsules
  Arms: CD-008-0045 40 mg/day; CD-008-0045 60 mg/day
Drug: Placebo — Placebo capsules
  Arms: CD-008-0045 40 mg/day; Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-finding pilot study to assess the efficacy and safety of CD-008-0045 in patients with Generalized Anxiety Disorder (GAD). Each patient will participate in the study for the period of approximately 10 weeks: Screening and Run-in period: 1 week; Study Treatment period: 8 weeks; Follow-up period: 1 week.

DETAILED DESCRIPTION:
The study drug CD-008-0045 has a multi-targeted activity, i.e., able to inhibit adrenergic, dopamine, serotonin, and histamine receptors, thus allowing to assume its wide therapeutic potential. At Screening, the patients who meet the inclusion/exclusion criteria will be included into one-week single-blind Placebo Run-in period. At Week 0 the patients will be randomized to receive CD-008-0045 60 mg daily, CD-008-0045 40 mg daily or Placebo for 8 weeks. The potential withdrawal syndrome will be assessed during one-week Follow-up Period.

ELIGIBILITY:
Inclusion criteria:

1. Signed Informed Consent Form;
2. Age 18 years and older;
3. Generalized anxiety disorder diagnosed according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria and International Classification of Diseases (ICD-10);
4. Hamilton Anxiety Rating Scale (HARS) values at Screening and on Randomization Visit (Week 0): Total score ≥ 20; Item 1 (Anxious mood) and Item 2 (Tension) scores ≥ 2;
5. The CGI-S score ≥ 4 (moderate severity and higher) at Screening and on Randomization visit (Week 0);
6. Consent of patients to use adequate contraception methods throughout the study. Adequate contraception methods include:

   * Condoms with spermicide for males;
   * For females (at their discretion):

     * oral contraceptives
     * condoms with spermicide (for the partner)
     * diaphragm with spermicide
     * cervical cap with spermicide
     * intrauterine device
7. Ability to comply with all Study Protocol requirements.

Exclusion criteria:

1. Pregnant or lactating women, or women planning to get pregnant during the clinical study; women of childbearing potential (including those without history of surgical sterilization and women with <2 years of post-menopause) not using adequate contraception methods;
2. Item 1 (Depressed mood) of the Hamilton Depression Rating Scale (HAMD) score ≥ 2;
3. Hamilton Depression Rating Scale (HAMD) total score > 13;
4. Confirmed diagnosis of depressive episode, recurrent depressive disorder, bipolar affective disorder in history or at Screening;
5. Confirmed diagnosis of schizophrenia in history or at Screening;
6. Confirmed diagnosis of panic disorder in history or at Screening;
7. Phobic anxiety disorders (agoraphobia, social phobia, unspecified phobic anxiety disorder) in history or at Screening;
8. Disorders of personality or behavior in history or at Screening;
9. Post-traumatic stress disorder diagnosed within 12 months prior to Screening;
10. Eating disorders diagnosed within 12 months prior to Screening;
11. Somatoform disorders in history or at Screening;
12. Obsessive-compulsive disorder in history or at Screening;
13. Epilepsy, seizures, head trauma with loss of consciousness, tumors, inflammatory, or demyelinating diseases of the central nervous system, stroke in history;
14. Pheochromocytoma;
15. Malignancies diagnosed within the last 5 years (except for the cured basal cell carcinoma);
16. Significant cardiovascular diseases diagnosed at present or within 12 months prior to Screening, including: Chronic heart failure, class III or IV (according to New York Heart Association classification); severe arrhythmia requiring treatment with class Ia, Ib, Ic, or III antiarrhythmic drugs; unstable angina; myocardial infarction; heart and coronary artery surgery; significant valvular heart disease; uncontrolled hypertension with systolic blood pressure > 180 mm Hg and diastolic blood pressure > 110 mm Hg; pulmonary embolism or deep vein thrombosis;
17. Nephrotic syndrome; moderate to severe chronic renal failure or significant renal diseases with creatinine level >1.5 mg/dL (132 μM/L) in males and > 1.4 mg/dL (123 μM/L) in females, or glomerular filtration rate (GFR) < 60 mL/min;
18. HIV, hepatitis B or C, liver cirrhosis in history; AST, ALT, or serum alkaline phosphatase ≥ 2.5 times above the upper limit of normal; total bilirubin level ≥ 2 times above the upper limit of normal at Screening;
19. Significant dysfunctions of the thyroid gland in decompensation stage;
20. Anemia (hemoglobin level ≤ 105 g/L in females or ≤ 115 g/L in males); significant blood loss, or collection of at least one volumetric unit of donated blood (≥ 500 ml), or blood transfusion within 12 weeks prior to Screening;
21. Any uncontrolled concomitant somatic disease, including that with a stable treatment regimen;
22. Drugs administered for generalized anxiety disorder, starting from Screening and throughout the study, including antidepressants, Pregabalin, benzodiazepines, antipsychotics;
23. Fluoxetine use within 21 days prior to Screening and throughout the study;
24. Known allergy, hypersensitivity or contraindications to CD-008-0045;
25. Electroconvulsive therapy within 3 months prior to Screening;
26. Psychotherapy within 3 months prior to Screening and/or at the time of enrollment into the study;
27. Use of prohibited drug therapy from the moment of Screening and throughout the study;
28. Administration of any study drug or participation in another clinical study within 3 months prior to Screening (except for cases when the patient was not administered the study drug during the study);
29. Addiction to tranquilizers or psychoactive substance abuse, including alcohol (history of episodic use is acceptable);
30. Inability to read or right; unwillingness to understand and comply with the Protocol procedures; non-compliance with drug dosage regimen or procedures which, in the Investigator's opinion, may affect the study results or the patient's safety and prevent the patient's participation in the study; any other concomitant diseases or severe mental disorders, which make the patient ineligible for participation in the study, limit the legal basis for Informed Consent procedure, or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment response | Baseline to Week 8
  Proportion of patients who demonstrate ≥ 50% decrease of the Hamilton Anxiety Rating Scale (HARS) [the values from 0 to 56; the higher scores mean a worse outcome] total score from baseline [% of patients]

SECONDARY OUTCOMES:
Change of the HARS total score | Baseline to Week 8, Week 8 to Week 9
  Mean change of HARS score [score]
Change in the score sum of the mental and somatic anxiety subscales of HARS | Baseline to Week 8
  Mean change of the score sum of the mental and somatic anxiety subscales of the HARS score [score]
Change of scores in items 1 (Anxious mood) and 2 (Tension) of HARS | Baseline to Week 8
  Mean change of the score in items 1 (Anxious mood) and 2 (Tension) of HARS [score]
Change of the sum of Hamilton Depression Rating Scale (HAM-D) scores | Baseline to Week 8, Week 8 to Week 9
  Mean change of HAM-D [the values from 0 to 52; the higher scores mean a worse outcome] score [score]
Change in the Clinical Global Impression - Severity Scale (CGI-S) | Baseline to Week 8, Week 8 to Week 9
  Mean change of CGI-S score [the values from 1 to 7; the higher scores mean a worse outcome] [score]
Clinical Global Impression - Improvement Scale (CGI-I) | Week 4, Week 8, Week 9
  Mean CGI-I score [the values from 1 to 7; the higher scores mean a worse outcome] [score]
Change of daytime somnolence level based on Visual Analogue Scale (VAS) | Baseline to Week 8, Week 8 to Week 9
  Mean change of VAS [the values from 0 to 10; the higher scores mean a worse outcome] score [score]
CD-008-0045 concentration prior to the next drug administration (Ctrough) | Week 4, Week 8
  Ctrough of CD-008-0045 [ng/ml]
M1 concentration prior to the next drug administration (Ctrough) | Week 4, Week 8
  Ctrough of M1 [ng/ml]
CD-008-0045 concentration 1 hour post drug administration (Cmax) | Week 4, Week 8
  Cmax of CD-008-0045 [ng/ml]
M1 concentration 1 hour post drug administration (Cmax) | Week 4, Week 8
  Cmax of M1 [ng/ml]
CYP2D6 polymorphism | Week 4
  CYP2D6 polymorphism [type of metabolism]
Incidence of adverse events (AE) and serious adverse events (SAE) | Baseline to Week 9
  Percent of patients with AEs and SAEs [% of patients]

CONTACTS AND LOCATIONS:
Overall Officials: Margarita A Morozova, MD,PhD,Prof, Principal Investigator — "Research Center for Mental Health" Scientific Institution
Locations (15):
- Russia (15):
  - Clinical Center LLC "Center for Psychotherapy "Support", Stavropol, Stavropol Kray
  - "Research Center for Mental Health" Scientific Institution, Moscow
  - Clinical Center LLC "University Headache Clinic", Moscow
  - Moscow Research Institute of Psychiatry "National Medical Research Center for Psychiatry and Narcology named after V.P. Serbsky", Moscow
  - Nizhny Novgorod Clinical Psychiatric Hospital No.1, Nizhny Novgorod
  - Clinical Center LLC "TREATMENT AND REHABILITATION RESEARCH CENTER "PHOENIX ", Rostov-on-Don
  - Ryazan Medical University, Department of Psychiatry, Ryazan
  - Clinical Center LLC "Doctor SAN", Saint Petersburg
  - Clinical Center LLC "Dynasty", Saint Petersburg
  - Leningrad Regional Psychoneurological Dispensary, Saint Petersburg
  - St. Petersburg "Psychoneurological dispensary #5", Saint Petersburg
  - Clinical Center LLC "LION-MED", Voronezh
  - Clinical Center LLC "Medical practice", Voronezh
  - Yaroslavl Regional Psychiatric Hospital, Yaroslavl
  - Clinical Center JSC "Medical Technologies", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No